CLINICAL TRIAL: NCT05105217
Title: Evaluation of Slit2 in Systemic Lupus Erythematosus and Systemic Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Safwat Mohamed, Resident doctor in Rhematology and rehabilitation department, Assiut University
Other Study IDs: Slit2 in SLE & SSC
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Slit2 biomarker — 1.Assessment of slit2 level in SLE patients and its correlation with disease activity.
  2-Assessment of slit2 level in SSC patients and its correlation with disease activity

SUMMARY:
1.Assessment of slit2 level in SLE patients and its correlation with disease activity.

2-Assessment of slit2 level in SSC patients and its correlation with disease activity

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is the most serologically and clinically diverse autoimmune disease. Immune dysregulation leads to excess production of autoantibodies and immune complexes. excess complement activation, and insidious tissue inflammation in patients with SLE.

SLE is characterized by multisystem involvement commonly affecting the skin, renal, and musculoskeletal systems .

Lupus nephritis is an important cause of both acute kidney injury and chronic kidney disease that can result in end-stage renal disease. Its pathogenic mechanisms are characterized by aberrant activation of both innate and adaptive immune responses, dysregulation of inflammatory signaling pathways, and increased cytokines production .

Systemic sclerosis (SSC) is an autoimmune disease with characteristic vascular damage and fibrosis of the skin and internal organs. Diagnosis of SSC is mainly based on the clinical course and features in addition to laboratory findings including autoantibody profiles

. Slit2, as a member of the Slit family, is secreted glycoprotein. Slit2 functions by binding to its transmembrane receptor Robo. Robo has four isoforms (Robo14). Slit2-Robo regulates cell functions, such as regulating leukocytes in chemotaxis and promoting endothelial cell migration and tube formation.

Slit2 might promote the pathogenesis of LN by affecting various cell dysfunction in addition to leukocyte infiltration.

In SSC, vascular involvement is a primary event characterized by vascular tone dysfunction and microcirculatory abnormalities. Many classes of guidance molecules, such as members of the secreted glycoproteins Slits and their Roundabout (Robo) receptors, play critical roles in angiogenesis. Among these, Robo1 and Robo4 are expressed in endothelial cells. .

ELIGIBILITY:
Inclusion Criteria:

1. Adult SLE Patients who fulfilled the 2019 EULAR/ACR Classification criteria for Systemic Lupus Erythematosus .
2. Adult SSC patients who fulfilled the 2013 EULAR / ACR for SSC

Exclusion Criteria:

* Individuals with other autoimmune diseases

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Adult SLE Patients
  2. Adult SSC patients
  3. Adult healthy control
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
measure the level of slit2 by ELISA in SLE patients | baseline
  determining level of Slit2 in patients with SLE and define its correlation with disease activity

SECONDARY OUTCOMES:
measure the level of slit2 by ELISA in SSC patients | baseline
  determining level of Slit2 in patients with SSC and define its correlation with disease activity

REFERENCES:
- See also: Slit2 is a potential biomarker for renal impairment in systemic lupus erythematosus — https://doi.org/10.1007/s10238-020-00664-x
- See also: A review of advances in the understanding of lupus nephritis pathogenesis as a basis for emerging therapies [version 1; peer review: 2 approved] — https://doi.org/10.12688/f1000research.22438.1